CLINICAL TRIAL: NCT00982085
Title: The Status of Asthma in the Korean Military Personnel
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Armed Forces Capital Hospital, Republic of Korea (Other Government)
Responsible Party: Sei Won Lee, Armed Forces Capital Hospital
Other Study IDs: Asthma Prevalence in ROK
Record Dates: First submitted 2009-09-21; First posted 2009-09-22 (Estimated); Last update posted 2009-09-22 (Estimated); Status verified 2009-09

CONDITIONS: Asthma
Keywords: Asthma; Allergic rhinitis; Military
MeSH Terms: conditions — Asthma; Rhinitis, Allergic

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Soldiers: Soldiers: The soldiers who respond the questionnaires

SUMMARY:
The aim of this study is to evaluate the status of allergic diseases in the Korean military personnel.

DETAILED DESCRIPTION:
ISAAC (International Study of Asthma and Allergies in CHildhood) questionnaires are sent to military personnel in the republic of Korea. Military personnel are randomly selected representative of the number of soldiers in each area. We perform methacholine provocation test and MAST for current wheezer after informed consents.

ELIGIBILITY:
Inclusion Criteria:

* Korean military personnel who can respond questionnaire

Exclusion Criteria:

* Person who refuse to participate in this study

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Korean Military personnel who resign in South Korea.
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-02 (Estimated); Study Completion 2010-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sang Min Lee, MD, Principal Investigator — Armed Forces Capital Hospital
Locations (1):
- Armed Forces Capital Hospital, Seongnam-si, Gyeonggi-do, South Korea